CLINICAL TRIAL: NCT04013789
Title: Comparison of Two Daily Disposable Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLD523-P001
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Refractive Ametropia; Myopia
Keywords: eye strain; eye fatigue
MeSH Terms: conditions — Myopia; Asthenopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DACP FreshTech, then DACP (Other): DACP FreshTech contact lenses worn first, followed by DACP contact lenses, as randomized. Each product was worn in both eyes for approximately 8 hours per day for 1 week with a new pair of lenses worn each day.
  Interventions: Device: DACP FreshTech contact lenses; Device: DACP contact lenses
- DACP, then DACP FreshTech (Other): DACP contact lenses worn first, followed by DACP FreshTech contact lenses, as randomized.. Each product was worn in both eyes for approximately 8 hours per day, for 1 week with a new pair of lenses worn each day.
  Interventions: Device: DACP FreshTech contact lenses; Device: DACP contact lenses

INTERVENTIONS:
Device: DACP FreshTech contact lenses — Nelfilcon A soft contact lenses with a modified lens design
  Other Names: DAILIES® AquaComfort PLUS® FreshTech
Device: DACP contact lenses — Nelfilcon A soft contact lenses
  Other Names: DAILIES® AquaComfort PLUS®

SUMMARY:
The purpose of this study was to compare the clinical performance of the new DAILIES® AquaComfort PLUS® FreshTech (DACP FreshTech) contact lenses to an already marketed daily disposable contact lens, DAILIES® AquaComfort PLUS® (DACP).

DETAILED DESCRIPTION:
Subjects attended 4 scheduled visits for an expected duration of participation of 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months of soft contact lens wearing experience;
* Wears habitual lenses at least 5 days per week and at least 8 hours per day;
* Uses digital devices (computer, tablet, and/or smart phone) for an average of 4 hours per day;
* Experiences eye fatigue at least once per week attributable to digital device use with habitual lenses;
* Is willing to NOT use rewetting/lubricating drops during the period of study product exposure;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Routinely sleeps in contact lenses;
* Known pregnancy at time of enrollment;
* Binocular vision issues or issues of eye alignment;
* Any eye infection, inflammation, disease or abnormality that contraindicates contact lens wear;
* Use of medications as specified in the protocol;
* Ocular surgery within the past 12 months;
* Other protocol-specified exclusion criteria may apply.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Project Lead, Study Director — Alcon Research
Locations (1):
- Alcon Investigative Site, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single investigative site in the United States.
Pre-assignment Details: Of the 79 enrolled subjects, 11 were screen failures and 1 withdrew prior to randomization. This reporting group includes all randomized subjects (67).
Period: First Wear Period (1 Week)
Arm/Group | DACP FreshTech, Then DACP | DACP, Then DACP FreshTech
Started | 33 | 34
Completed | 33 | 34
Not Completed | 0 | 0
Period: Second Wear Period (1 Week)
Arm/Group | DACP FreshTech, Then DACP | DACP, Then DACP FreshTech
Started | 32 (One subject withdrew from the study between the first wear period and the second wear period.) | 34
Completed | 32 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects.
Groups:
- Overall: DACP FreshTech contact lenses and DACP contact lenses worn during Period 1 and Period 2 in a crossover assignment, as randomized.
Arm/Group | Overall
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 54
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Distance Visual Acuity (VA) With Study Lenses
Description: VA was assessed at a distance of 4 meters using a letter chart and was measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity.
Time Frame: Week 1, each product
Population: Full Analysis Set: All randomized subjects (as randomized) who were exposed to any study lenses, not including the optimized habitual and trial fit lenses.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- DACP FreshTech: DACP FreshTech contact lenses worn in both eyes for approximately 8 hours per day for 1 week with a new pair of lenses worn each day
- DACP: DACP contact lenses worn in both eyes for approximately 8 hours per day for 1 week with a new pair of lenses worn each day
Arm/Group | DACP FreshTech | DACP
Number analyzed (Participants) | 66 | 66
logMAR | -0.20 (0.06) | -0.22 (0.05)
Statistical Analysis 1: Comparison: DACP FreshTech vs DACP; Test type: Non-Inferiority — The noninferiority margin was set at 0.05; Mixed Effects Repeated Measures Model; Least Squares Mean Difference = 0.02, 95% CI 1-sided [upper limit 0.03], Standard Error of Mean 0.006 — DACP FreshTech minus DACP

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent to study exit, approximately 3 weeks. The safety analysis set included all all randomized subjects (as treated) who were exposed to any study lenses, not including the optimized habitual and trial-fit lenses.
Description: Adverse events (AEs) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects.
Groups:
- DACP FreshTech - Ocular; DACP FreshTech - Systemic / Nonocular: Nelfilcon A soft contact lenses with a modified lens design worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for approximately 7 days with a new pair of lenses worn each day.
- DACP - Ocular; DACP - Systemic / Nonocular: Nelfilcon A soft contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for approximately 7 days with a new pair of lenses worn each day.
Arm/Group | DACP FreshTech - Ocular | DACP FreshTech - Systemic / Nonocular | DACP - Ocular | DACP - Systemic / Nonocular
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/67 | 0/132 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/67 | 0/132 | 0/66
Other Adverse Events (participants affected / at risk) | 0/134 | 0/67 | 0/132 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT04013789/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT04013789/SAP_001.pdf